CLINICAL TRIAL: NCT05147168
Title: Quality of Life of Pancreatic Cancer Patients:Psychometric Validation of Chinese Version of the EORTC QLQ-PAN26 and EORTC QLQ-C30 in Taiwan
Brief Title: Quality of Life of Pancreatic Cancer Patients:Psychometric Validation of Chinese Version in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-11-012BC
Record Dates: First submitted 2021-11-22; First posted 2021-12-07 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer
Keywords: Quality of life; Psychometric Validation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Psychometric Validation of Chinese Version of the EORTC QLQ-PAN26 and EORTC QLQ-C30 in Taiwan

SUMMARY:
This study will investigate the reliability and validity of Chinese version of the quality of life scale in EORTC QLQ-PAN26 and EORTC QLQ-C30 on pancreatic cancer patients in Taiwan

DETAILED DESCRIPTION:
1. Verify the reliability and validity of Chinese version of the EORTC QLQ-C30 Quality of Life Scale and the chinese version of the EORTC QLQ-PAN26 Quality of Life Scale.
2. Verify the construct validity of the Chinese version of the EORTC QLQ-PAN26 Quality of Life Scale, perform factor analysis, test-retest reliability, and known group validity
3. Verify the criterion related validity of Chinese version of the EORTC QLQ-C30 Quality of Life Scale and the SF-36 Quality of Life Scale

ELIGIBILITY:
Inclusion Criteria:

1. Paitent who aged over 20, with clear consciousness, is capable of communicating with Chinese.
2. Pancreatic Cancer patients(stage I.II.III.IV)
3. The subject who agrees and is willing to participate in the research after explaining the purpose of the research.

Exclusion Criteria:

1. Patient who is younger than 20 years old, illiterate, or is unable to cooperate with intervention measures.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic Cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2024-11-22 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (EORTC QLQ-C30 ) | baseline
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-C30 consists three subscales with 30 questions.The EORTC QLQ-C30 included three subscales: functioning scales (15questions), symptom scales (13 questions), and global health status (2questions). The reliability and validity of Cronbach'α was 0.52-0.89. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | baseline
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | 2nd or 3rd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life(SF-36) | baseline
  This scale was evaluated by self-assessment of various clinical problems for a month.The SF-36 included eight subscales.The reliability and validity of Cronbach'α was 0.57.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Study Chair — National Taipei University of Nursing and Health Sciences
Locations (1):
- Taipei Veterans General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and receive the authors consent